CLINICAL TRIAL: NCT06133569
Title: A Multicenter, Waitlist Controlled, Randomized Clinical Trial of the Effectiveness of a Self Help Program Based on Cognitive Behavioral Therapy for Individuals with Sexual Interest in Children.
Brief Title: ReDirection - Self Help Program for Individuals with Sexual Interest in Children
Acronym: ReDirection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Centre for Psychiatry Research, Region Stockholm, Sweden (Unknown); Linkoeping University (Other Government); Universitat Jaume I, Spain (Unknown); Protect Children Organisation, Finland (Unknown); National Institute of Mental Health, Czech Republic (Other); Academy of the Police Force, Bratislava, Slovakia (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Christoffer Rahm, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02321-01; 101084355-BRIDGE-ISF-2021 (Other: European Commission)
Record Dates: First submitted 2023-10-12; First posted 2023-11-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Child Abuse Sexual; Pedophilia
Keywords: Child sexual abuse material; Cognitive behavioral therapy; Internet based self-help program; Individuals with sexual interest in children
MeSH Terms: conditions — Pedophilia

STUDY DESIGN:
Intervention Model Description: Participants are allocated to either the ReDirection intervention or waitlist during the initial phase of the study and those who receive waitlist receive ReDirection during the second phase of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ReDirection (Experimental): ReDirection is a self help program based on cognitive behavioral therapy methodology and consists of five modules. The program aims to help participants reduce their CSAM use by gaining a better understanding of, and skills to manage risky sexual thoughts, feelings, and behaviors.
  Interventions: Behavioral: ReDirection
- Waitlist (No Intervention): Participants are on a waitlist which means they have no active intervention, only weekly measurements with the same questionnaires as in the active arm.

INTERVENTIONS:
Behavioral: ReDirection — Self help program based on principles for cognitive behavioral therapy
  Arms: ReDirection

SUMMARY:
The overall aim of the study is to evaluate the effectiveness of the ReDirection program for individuals with low or medium risk to commit child sexual abuse.

Primary question: Is ReDirection a feasible, effective, and safe method in reducing low to medium risk participants' use of CSAM and related behaviors?

DETAILED DESCRIPTION:
The present research project aims to contribute to the further development of accessible, evidence-based and safe care for people with concerns about their sexual interest regarding children, and that are using child sexual abuse material (CSAM), so that these people can access treatment according to their needs and level of risk, with the objective of reducing the risk for child sexual abuse and improving the health of the group.

More concretely, we aim to evaluate a revised version of an already available cognitive-behavioral self-help program, ReDirection, with the aim of testing whether this intervention can reduce sexual interest regarding children and CSAM use, in a group of people assessed as being at low or medium risk of committing sexual abuse of children. The intervention will be available in seven languages and will be tested in six countries.

Primary research question: Is ReDirection a feasible, effective, and safe method in reducing low to medium risk participants' use of CSAM and related behaviors?

Secondary research questions: Is ReDirection effective in reducing research subjects' overall risk of committing sexual acts involving children? Does ReDirection reduce specific dynamic risk factors for committing CSA?

ReDirection is based on cognitive behavioral therapy and consists of five modules. The program aims to help participants reduce their CSAM use by gaining a better understanding of, and skills to manage risky sexual thoughts, feelings, and behaviors. At the end of the program, participants are offered an anonymous follow-up chat and if needed during the program, participants can contact a practitioner via chat.

Research subjects will be recruited through Darknet and Clearnet. Darknet refers to websites that are accessible via TOR or similar services. The interventions are provided by practitioners and researchers in the relevant countries.

ReDirection will be evaluated through an international multicenter study using randomized wait-list controlled design.

The research subjects will sign a written consent form on the Iterapi platform without disclosing personal data such as name or location. During the subsequent screening interview via chat or voice call on Iterapi, participation criteria are ensured, questions are answered, and the consent to participate is confirmed. The research subjects are thus admitted to the study.

After inclusion, participants answer the baseline survey which consists of validated self-assessment questionnaires with both multiple choice and free-text answers.

Weekly during, after the waitlist, and after the therapeutic intervention, research subjects answer questions to evaluate the effectiveness and safety of the interventions.

A Statistical Analysis Plan (SAP) based on pilot study is pre-registered at the OSF platform. The SAP describes sample size calculations, and planned analyses of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient language skills: English, Swedish, Finnish, Czech, Slovak, German, or Spanish
* concern about sexual interest regarding children*,
* CSAM use past six month
* Low to medium risk for committing child sexual abuse according to the SChiMRA scale

Exclusion Criteria:

- Participants with a severe psychiatric illness (such as high acute suicide risk or severe substance abuse) will be excluded, or lack of serious intentions to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Sexual interest involving children | Pre-intervention, during the intervention, and immediately after the intervention.
  Measured by Sexual Symptom Assessment Scale (SASS)(0-48 points; higher scores indicate more interest).
Child sexual abuse material usage | Pre-intervention, during the intervention, and immediately after the intervention.
  Measured with Sexual Child Molestation Risk Assessment (SChiMRA+), part B, item 1 (self-reported time spent last week in hours watching CSAM) including 3 follow up questions (about time/day, severity, and of youngest child).
Other behaviors related to sexual interest in children. | Pre-intervention, during the intervention, and immediately after the intervention.
  Time spent last week (hours), as self reported on the SChiMRA+ scale part B, item 4.
Depressive symtoms | Pre-intervention, and immediately after the intervention.
  Scores on the PHQ-9 questionnaire (Patient Health Questionnaire; 0-27 points; higher scores indicate more severe depressive symptoms).

SECONDARY OUTCOMES:
Dynamic risk for committing child sexual abuse | Pre-intervention, during the intervention,and immediately after the intervention.
  Scores on Acute-2007 (21 items; 0-42 points; higher scores indicate higher dynamic risk for committing child sexual abuse)
Level of hypersexuality | Pre-intervention, and immediately after the intervention.
  Scores on the HBI-19 questionnaire (Hypersexual Behavior Inventory; 19-95 points; higher scores indicate higher level of sexuality; more than 52 points indicate hypersexuality)

CONTACTS AND LOCATIONS:
Locations (6):
- National Institute of Mental Health, Klecany, Czechia
- Protect Children NGO, Helsinki, Finland
- [University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Bratislava Police Academy, Bratislava, Slovakia
- Universitat Jaume I, Castelló, Spain
- Centre for psychiatry research, Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Web page for the study — https://www.iterapi.se/sites/bridge